CLINICAL TRIAL: NCT04817696
Title: Epidemiology of Chronic Pain as Part of Post-resuscitation Syndrome. Multicenter Prospective Non-interventional Study
Brief Title: Epidemiology of Chronic Pain as Part of the Post-intensive Care Syndrome
Acronym: ALGO-REA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0020
Record Dates: First submitted 2021-02-01; First posted 2021-03-26 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Critical Care; Chronic Pain
Keywords: PICS; Post Intensive Care Syndrome; Chronic Pain; Critical Care
MeSH Terms: conditions — Chronic Pain; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients without chronic pain symptoms — Verbal score < 3 at 3 months
Other: Patients with chronic pain symptoms — Verbal score ≥ 3 at 3 months

SUMMARY:
Post-intensive care syndrome is an entity of cognitive, physical and mental health disorders occurring and persisting after ICU discharge and responsible of disabilities and decrease of quality of life. Nowadays mental and cognitive health impairments appear to be well known but few data are available about chronic pain after a critical care illness. The aim of the study is to determine the incidence and the risks factors of chronic pain after ICU.

DETAILED DESCRIPTION:
Post-intensive care syndrome is receiving growing interest because of the chronic health issues secondary to a critical care admission: neurocognitive impairment, motor sequelae, mood disturbances. These chronic health issues bear tremendous burden for patients and next-of-kin. Among these chronic health issues, chronic pain symptoms could have major consequences on the patient's quality of life. In the local single-center follow-up experience, 6 months after a patient's admission in the critical care unit, around 20% of patients displayed chronic pain symptoms. The investigators have addressed these patients to pain care specialists, with successful treatment success. However, the evaluation of pain symptoms remains simplistic; moreover, the incidence of chronic pain symptoms in patients after critical care unit admission, receives little attention in the literature although these symptoms may literally blunt out all other health issues. The incidence and type of chronic pain symptoms has been poorly described, to the best of knowledge.

The aim of this study is to perform a multi-center nationwide epidemiologic study of chronic pain symptoms after a critical care unit admission. The investigators intend to describe the incidence of chronic pain assessed with a Simple Verbal Score ≥ 3, 3 months after the ICU admission. The investigators also intend to describe the incidence of painful symptoms, at ICU discharge as well as the type of pain symptoms (ie neuropathic pain) at discharge and at 3 months using the ID-Pain scale. The evaluation at 3 months will be performed during a physical follow-up or self-assessed by the patient. The investigators intend to explore the risk factors associated with chronic pain, as an exploratory analysis.

The investigators are performing a nation-wide multicentric study. At this point 24 centers are participating to this study and the investigators expect to include 700 patients with a 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria :

* All patients admitted in ICU
* ICU length-of-stay ≥ 48 hours
* No major cognitive impairment that could prevent pain evaluation

Exclusion Criteria :

* Patient under 18-year-old
* Patient under guardianship
* Patient unable to communicate or quantify pain with a Verbal Score and ID-Pain score
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in ICU with a length of stay > 48 hours and without major cognitive impairment that could prevent an accurate evaluation of pain
Sampling Method: Non-Probability Sample
Enrollment: 1079 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Presence of pain (Simple Verbal Scale ≥3) persisting at 3 months after ICU admission | 3 months after the ICU admission
  Chronic pain is defined as a Simple Verbal Scale (ranging from 0 - no symptoms- to 10 - worst symptoms imaginable-) ≥ 3.

SECONDARY OUTCOMES:
Intensity of pain, and risk factors associated with pain at 3 months after ICU admission | ICU discharge (median 7 days)
  The incidence of pain defined as a Simple Verbal Scale (ranging from 0 - no symptoms- to 10 - worst symptoms imaginable-) ≥ 3
Type of pain (ie neuropathic) | ICU discharge (median 7 days) and at 3 months after admission
  The Type of pain will be assessed with the score ID-Pain at ICU discharge, and 3 months after discharge. The ID-Pain is a 6-item scores that characterizes pain.The score ranges from 0 to 5. A score of 2-3 is predictive of a probable neuropathic pain and a score of 4-5 is highly associated with a neuropathic pain. Pain assessment tools require an auto-evaluation, performed by the patient
Pain management and risk factors in the ICU (Use of Remifentanyl) | Median 7 days
  Binary information (yes/no)
Pain management and risk factors in the ICU (Use of continuous intra-venous Morphine) | Median 7 days
  Binary information (yes/no)
Pain management and risk factors in the ICU (Use of continuous intra-venous Ketamine) | Median 7 days
  Binary information (yes/no).
Pain management and risk factors in the ICU (Use of anti-hyperalgesia medication (ie : anti-epileptique drugs, gabapentine, tricyclic anti-depressive drugs)) | Median 7 days
  Binary information (yes/no).
Pain management and risk factors in the ICU (Use of locoregional anesthesia) | Median 7 days
  Binary information (yes/no).
Pain management and risk factors in the ICU (Type surgery and invasive procedures during ICU: Neurosurgery, orthopedic surgery spine surgery, abdominal surgery, thoracic surgery, thoracic drain) | Median 7 days
  Binary information (yes/no)
Pain management and risk factors in the ICU | Median 7 days
  • These outcomes and measures will be analyzed separately in the regression multivariable models of chronic pain and neuropathic pain.
Demographic data | Baseline
  * Age
  * Sex
  * SAPS II
  * Type of ICU admission
  * Chronic Cardiovascular diseases: ischemic cardiomyopathy, hypertention
  * Chronic use of pain killers
General ICU data (Length of invasive mechanical ventilation) | ICU discharge (median 7 days)
  Measured as the number of days between succesfull weaning of mechanical ventilation and initiation. Median duration : 7 days
General ICU data | ICU discharge (median 7 days)
  • ARDS. Defined as a PaO2/FiO2 ratio < 300mmHg, according to the Berlin definition (JAMA 2012). Binary information (yes/no). Median duration of monitoring : 7 days
General ICU data ( Use of prone positionning during invasive mechanical ventilation) | ICU discharge (median 7 days)
  Binary information (yes/no). Median duration of monitoring :7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourdiol A, Legros V, Vardon-Bounes F, Rimmele T, Abraham P, Hoffmann C, Dahyot-Fizelier C, Jonas M, Bouju P, Cirenei C, Launey Y, Le Gac G, Boubeche S, Lamarche E, Huet O, Bezu L, Darrieussecq J, Szczot M, Delbove A, Schmitt J, Lasocki S, Auchabie J, Petit L, Kuhn-Bougouin E, Asehnoune K, Ingles H, Roquilly A, Cinotti R; ALGO-REA study group; Atlanrea Group; Societe Francaise d'Anesthesie-Reanimation-SFAR Research Network. Prevalence and risk factors of significant persistent pain symptoms after critical care illness: a prospective multicentric study. Crit Care. 2023 May 25;27(1):199. doi: 10.1186/s13054-023-04491-w. PMID 37226261